CLINICAL TRIAL: NCT06457425
Title: An Open-Label, Positive Drug-Controlled, Parallel, Multicenter Phase II Clinical Trial of the Efficacy, Safety, and Pharmacokinetics of Flonoltinib Maleate Tablets in Patients With Intermediate to High-Risk Myelofibrosis
Brief Title: A Phase II Clinical Trial of Flonoltinib Maleate Tablet in Intermediate-High Risk Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMF-02
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: MF,PMF,PPV-MF,PET-MF
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low dose group (Experimental): Flonoltinib 50mg
  Interventions: Drug: Flonoltinib 50mg
- high dose group (Experimental): Flonoltinib 100mg
  Interventions: Drug: Flonoltinib 100mg
- control group (Active Comparator): Ruxolitinib
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Flonoltinib 50mg — Flonoltinib 50mg, QD
  Arms: low dose group
Drug: Flonoltinib 100mg — Flonoltinib 100mg, QD
  Arms: high dose group
Drug: Ruxolitinib — For patients with platelet counts between 100×10^9/L and 200×10^9/L, the recommended starting dose is 15 mg twice daily (bid). For patients with platelet counts >200×10^9/L, the recommended starting dose is 20 mg bid. For patients with platelet counts between 50×10^9/L and <100×10^9/L, the recommended maximum starting dose is 5 mg bid.
  Arms: control group

SUMMARY:
This trial adopts a multicenter, open-label, positive drug parallel control clinical trial design, planning to enroll approximately 75 MF participants. Eligible participants will be stratified and assigned in a 1:1:1 ratio to the low-dose flonoltinib maleate tablet group, high-dose flonoltinib maleate tablet group, or the ruxolitinib tablet group. Stratification factor include the Dynamic International Prognostic Scoring System (DIPSS) risk classification (intermediate-2 and high risk)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restrictions;
2. Diagnosed with primary myelofibrosis (PMF) according to WHO criteria (2016 edition) or post-polycythemia vera myelofibrosis (PPV-MF) or post-essential thrombocythemia myelofibrosis (PET-MF) according to IWG-MRT criteria;
3. Evaluated as intermediate-2 or high-risk myelofibrosis according to the Dynamic International Prognostic Scoring System (DIPSS) risk classification;
4. Expected survival ≥ 24 weeks;
5. ECOG score of 0-2;
6. Splenomegaly: palpable spleen edge reaching or exceeding 5 cm below the costal margin (distance from the intersection of the left midclavicular line and the left costal margin to the farthest point of the spleen); or not palpable due to body habitus (obesity) but confirmed by magnetic resonance imaging (MRI ) (or CT scan if necessary) at screening with spleen volume ≥ 450 cm³;
7. Blasts in peripheral blood and bone marrow ≤ 10%; 8) Within 7 days before the first dose, absolute absolute neutrophil count (ANC )≥ 1.0×10^9/L, platelet count ≥ 50×10^9/L, hemoglobin (HGB )> 60 g/L (participants should not have received growth factors, colony-stimulating factors, thrombopoietic agents, or platelet transfusions within 2 weeks before the baseline assessment prior to the first dose); 9) Major organ function basically normal within 7 days before the first dose; 10) Able to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Previous anticancer treatment-related toxic reactions have not recovered to grade 1 or below (excluding alopecia and conditions specified in inclusion criteria 8 and 9), or have not fully recovered from previous surgery (major surgery within 4 weeks);
2. Hypersensitivity, allergic to the investigational drug or its excipients;
3. Previous intolerance or resistance to ruxolitinib;
4. Use of JAK inhibitors within 4 weeks before the first dose;
5. Any significant clinical and laboratory abnormalities that, in the investigator's opinion, affect safety evaluation;
6. History of congestive heart failure, unstable angina, myocardial infarction, cerebrovascular accident (excluding lacunar infarction), or pulmonary embolism within 6 months prior to screening;
7. Impaired cardiac function or arrhythmic disease requiring treatment at screening;
8. Any active infection requiring intravenous antibiotic treatment at screening;
9. Active tuberculosis infection within 48 weeks prior to screening or latent tuberculosis infection indicated by tuberculosis-related tests during the screening period;
10. Patients who have undergone splenectomy or received radiation therapy to the spleen area within 12 months before the first dose;
11. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, except for: a) HBV infection: Patients with positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) with undetectable peripheral blood HBV-DNA (below the detection limit of the testing laboratory) can be enrolled; they must continue antiviral therapy and have HBV-DNA testing every 12 weeks and at the end of treatment (EOT); b) HCV seropositive patients with negative HCV RNA can be enrolled.
12. Positive for human immunodeficiency virus antibody (HIV-Ab) or Treponema pallidum antibody (TP-Ab) (patients with positive Treponema pallidum antibody can have a titer test, and the investigator will determine eligibility based on comprehensive judgment);
13. Patients with epilepsy or those using psychiatric drugs or sedatives at screening (excluding those used for sleep purposes);
14. Pregnant or breastfeeding women, and patients with reproductive potential (male and female) who refuse to use contraceptive measures during the trial and for 6 months after the trial;
15. Patients who have had another malignancy within 5 years before the first dose (excluding cured in-situ carcinoma and basal cell carcinoma of the skin);
16. Patients with other severe diseases that, in the investigator's opinion, may affect safety or compliance;
17. Patients who participated in other clinical trials of investigational drugs or medical devices within 1 month before the first dose and used the investigational drug or device;
18. Use of any treatment for MF (other than JAK inhibitors) within 2 weeks or 5 half-lives (whichever is longer) before the first dose, any immunomodulatory agents (e.g., thalidomide), any immunosuppressants, ≥10 mg/day prednisone or equivalent biological potency corticosteroids, or growth factors (e.g., erythropoietin (EPO)) (Traditional Chinese medicine should be stopped 1 day before the first dose);
19. Patients with a history of congenital or acquired bleeding disorders;
20. Other factors that the investigator deems unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with ≥35% reduction in spleen volume from baseline(Evaluation by IRC) | Week 24
  Percentage of subjects with ≥35% reduction in spleen volume from baseline(Evaluation by IRC)

SECONDARY OUTCOMES:
Percentage of subjects with ≥35% reduction in spleen volume from baseline (Evaluation by researcher) | Week 24
  Percentage of subjects with ≥35% reduction in spleen volume from baseline(Evaluation by researcher)
Percentage of subjects with ≥35% reduction in spleen volume from baseline (Evaluation by researcher) | Week 12
  Percentage of subjects with ≥35% reduction in spleen volume from baseline (Evaluation by researcher)
Percentage of subjects with ≥35% reduction in spleen volume from baseline (Evaluation by IRC) | Week 12
  Percentage of subjects with ≥35% reduction in spleen volume from baseline( Evaluation by IRC)
Percentage of subjects with ≥50% reduction in MPN-SAF TSS scale total symptom score | Week 24 and Week 12
  Percentage of subjects with ≥50% reduction in MPN-SAF TSS scale total symptom score
Objective response rate (ORR = CR + PR) per the IWG-MRT consensus criteria. | Week 24
  Objective response rate (ORR = CR + PR) per the IWG-MRT consensus criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Xiao, Doctor, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences; Ting Niu, Doctor, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality